CLINICAL TRIAL: NCT07122622
Title: Role of 2D-shear Wave Spleen Elastography in Assessing Clinically Significant Portal Hypertension and High-risk Varices in Patients With Advanced Compensated Chronic Liver Disease.
Brief Title: 2D-shear Wave Spleen Elastography in Clinically Significant Portal Hypertension and High-risk Varices
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Garcovich Matteo, Doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 7514
Record Dates: First submitted 2025-06-02; First posted 2025-08-14 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Portal Hypertension Related to Cirrhosis; Esophageal Varices
MeSH Terms: conditions — Esophageal and Gastric Varices

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to evaluate the role of spleen shear wave elastography (SWE-SSM) for ruling in and ruling out clinically significant portal hypertension (CSPH) in patients with compensated advanced chronic liver disease (cACLD) and for ruling in and ruling out high-risk esophageal varices (HRV) in patients with CSPH. Secondary objectives of the study include the investigation of the correlation between SWE-SSM and portal pressure in a subgroup of patients undergoing hepatic venous pressure gradient (HVPG) measurement and between SWE-SSM and transient elastography (TE-SSM).

The values of SWE-SSM and SWE-LSM will be assessed during the ultrasound examination to which the patient will be subjected according to their care pathway. If inclusion criteria are met and informed consent is obtained, spleen elastography will be carried out (in addition to the routine SWE-LSM planned in clinical practice). Spleen elastography will not alter the standard ultrasound examination but represents a non-invasive diagnostic addition.

There will be no treatment or experimental intervention that will modify the patient's condition or directly influence their clinical course. The aim is to collect data based on clinical observations without altering the treatment or the natural course of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years;
* SWE-LSM ≥9 kPa and/or TE-LSM ≥15 kPa;

Exclusion Criteria:

* Presence of transjugular intrahepatic porto-systemic shunt (TIPS);·
* Surgical absence of the spleen;
* Grade 3 ascites;
* History of variceal bleeding;
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referring to the Diagnostic and Interventional Ultrasound UOSD of the digestive system disease center of the University Hospital Policlinico A.Gemelli of Rome to undergo an ultrasound of the upper abdomen as part of their clinical pathway.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2027-08-20 (Estimated); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
CSPH | 2 years
  The following data will be collected:
  * Shear Wave Elastography of the spleen (SWE-SSM): continuous variable, expression of splenic stiffness, measured in kPa;
  * Shear Wave Elastography of the liver (SWE-LSM): continuous variable, expression of hepatic stiffness, measured in kPa;
  * Transient Elastography of the spleen (TE-SSM): continuous variable, expression of splenic stiffness, measured in kPa;
  * Transient Elastography of the liver (TE-LSM): continuous variable, expression of hepatic stiffness, measured in kPa;
  * Bipolar diameter of the spleen: measured in centimeters
  * Ascites yes/no;
  * Collateral circulation yes/no;
  * Encephalopathy yes/no;
  * Non selective beta-blockers yes/no;
  * Hepatic Venous Pressure Gradient (HVPG): continuous variable, portosystemic pressure gradient, measured in mmHg.

SECONDARY OUTCOMES:
HRV | 2 years
  The following data will be collected:
  * Shear Wave Elastography of the spleen (SWE-SSM): continuous variable, expression of splenic stiffness, measured in kPa;
  * Shear Wave Elastography of the liver (SWE-LSM): continuous variable, expression of hepatic stiffness, measured in kPa;
  * Transient Elastography of the spleen (TE-SSM): continuous variable, expression of splenic stiffness, measured in kPa;
  * Transient Elastography of the liver (TE-LSM): continuous variable, expression of hepatic stiffness, measured in kPa;
  * Bipolar diameter of the spleen: measured in centimeters
  * Endoscopic data: esophageal varices classified as F1, F2, F3 and with/without red spots.

CONTACTS AND LOCATIONS:
Locations (1):
- Ultrasound diagnostic and interventional service "Policlinico A.Gemelli", Roma, Italia, Italy